CLINICAL TRIAL: NCT00312026
Title: A Phase IV Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of 1.0 mg/kg Efalizumab in Adult Patients With Moderate to Severe Plaque Psoriasis Involving the Hands and/or Feet
Brief Title: A Study to Evaluate the Safety and Efficacy of Efalizumab in Adult Patients With Plaque Psoriasis Involving the Hands and/or Feet
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACD3753g
Record Dates: First submitted 2006-04-05; First posted 2006-04-07 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Psoriasis
Keywords: Plaque Psoriasis; Hands; Feet; Hand
MeSH Terms: conditions — Psoriasis | interventions — efalizumab

INTERVENTIONS:
Drug: efalizumab

SUMMARY:
This is a Phase IV randomized, double-blind, placebo-controlled study to evaluate the safety and efficacy of SC efalizumab in adult patients (18 years of age and older) with chronic moderate to severe plaque psoriasis involving the hands and/or feet who have had no previous exposure to efalizumab. The study will consist of a screening period, a treatment period, and an observation period.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent and Health Insurance Portability and Accountability Act of 1996 (HIPAA) documents
* Be aged 18 years or older
* Have chronic (6 months or greater) moderate to severe plaque psoriasis involving the hands and/or feet with or without pustules and with or without psoriasis at other sites
* Have a PGA rating of moderate (3) or severe (4) for hand and/or foot psoriasis
* Be a candidate for systemic therapy in the opinion of the investigator
* Be naive to efalizumab treatment
* Weigh no more than 125 kg
* For women of childbearing potential, use a method of contraception acceptable to the investigator to prevent pregnancy and agree to continue to practice an acceptable method of contraception for the duration of their participation in the study and for 6 weeks after the last dose of efalizumab

Exclusion Criteria:

* Have a history of hypersensitivity to efalizumab or any of its components
* Are using any excluded therapy
* Have a history of or ongoing alcohol or illegal drug abuse
* Have a history of or an ongoing uncontrolled serious bacterial, viral, fungal, or atypical mycobacterial infection. This includes diagnoses that required more than 2 weeks of therapy, such as endocarditis and osteomyelitis, that have been treated in the past 6 months. In addition, if the patient is currently receiving antibiotics, antivirals, or antifungals for an infection or for suppression or prophylaxis for any diagnosis, the patient will be excluded.
* Have any history of opportunistic infections (e.g., systemic fungal infections, parasites)
* Are seropositive for hepatitis B antigen, hepatitis C antibody, or human immunodeficiency virus (HIV). Patients will undergo testing during screening, and any patients who are seropositive for hepatitis B antigen, hepatitis C antibody, or HIV will be excluded.
* Have a history of active tuberculosis or are currently undergoing treatment for tuberculosis. A purified protein derivative (PPD) test or chest x-ray will be performed at the screening visit. Patients with a positive PPD test (not due to BCG vaccination) or chest x-ray will be excluded.
* Have the presence or history of malignancy within the past 5 years, including lymphoproliferative disorders. Patients with a history of fully resolved basal or squamous cell skin cancer may be enrolled.
* Are pregnant or lactating women
* Have a diagnosis of hepatic cirrhosis, regardless of cause or severity
* Have a history of thrombocytopenia
* Have a history of hemolytic anemia
* Have a history of clinically significant anemia
* Have a WBC count <4,000 cells/uL or >14,000 cells/uL
* Have a hematocrit (HCT) <30% or a hemoglobin (Hgb) level <11 g/dL
* Have a platelet count <150,000 cells/uL
* Have hepatic enzyme levels ≥3 times the upper limit of normal
* Have a serum creatinine level ≥2 times the upper limit of normal
* Have been exposed to any experimental drugs or treatments within 30 days or 5 half-lives, whichever is longer, prior to the screening visit
* Have had any previous exposure to efalizumab
* Have been vaccinated with a live virus or live bacteria within the 14 days prior to the first dose of efalizumab
* Have any medical condition that, in the judgment of the investigator, would jeopardize the patient's safety following exposure to study drug (efalizumab or placebo equivalent) or would significantly interfere with the patient's ability to comply with the provisions of this protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75
Dates: Start 2006-03-30; Primary Completion 2006-11-28 (Actual); Study Completion 2006-11-28 (Actual)

PRIMARY OUTCOMES:
The primary efficacy outcome measure is the proportion of patients who achieve a PGA rating of clear (0), almost clear (1), or mild (2) at Day 84.

SECONDARY OUTCOMES:
The proportion of patients who achieve a PGA rating of clear (0), almost clear (1), or mild (2) at Day 42
The proportion of patients who achieve a PGA rating of clear (0) or almost clear (1) at Day 84
The change from Day 0 to Day 84 in the following PRO measures: SF 36, PDS, Work Loss Questionnaire
The change from Day 0 in PGA rating (i.e., the number of categories changed) at Day 84

CONTACTS AND LOCATIONS:
Overall Officials: Ivor Caro, M.D., Study Director — Genentech, Inc.